CLINICAL TRIAL: NCT00717925
Title: A Phase 1 Study Of CMC-544 Administered As A Single Agent In Subjects With B-Cell Non-Hodgkin's Lymphoma
Brief Title: Study Evaluating Safety and Tolerability of Inotuzumab Ozogamicin (CMC-544) in Japanese Patients With B-cell Non-Hodgkin's Lymphoma (NHL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3129K1-103
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Lymphoma, B-Cell
Keywords: B-cell Non-Hodgkin's Lymphoma; NHL
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Inotuzumab Ozogamicin (CMC-544)

INTERVENTIONS:
Drug: Inotuzumab Ozogamicin (CMC-544) — Intravenous (IV) infusion, 1.3 - 1.8 mg/m2, every 28 days, 4 cycles

SUMMARY:
To assess the tolerability and the initial safety profile of Inotuzumab Ozogamicin (CMC-544) in patients with B-Cell Non-Hodgkin's Lymphoma (NHL).

ELIGIBILITY:
Inclusion Criteria:

* CD22-positive, B-cell NHL which has progressed after 1 or 2 prior therapies.
* Patients who have progressed after at least 1 prior chemotherapy regimen for indolent lymphoma, or 1/ 2 chemotherapy regimens, which include anthracylin or anthraquinon for aggressive lymphoma.
* Eastern Cooperative Oncology Group (ECOG) performance status: 0/ 1.

Exclusion Criteria:

* Patients must not have received monoclonal antibodies or radioimmunoconjugates within 3 months before first dose of test article.
* Patients must not have received bilateral pelvic irradiation.
* Patients must not have received chemotherapy, cancer immunosuppressive therapy, growth factors (except erythropoietin), or investigational agents within 4 weeks before first dose of test article.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events, dose-limiting toxicities, and changes in laboratory test results. | 4 months

SECONDARY OUTCOMES:
Tumor response (according to the International Response Criteria for Non-Hodgkin's Lymphomas). | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] Ogura M, Tobinai K, Hatake K, Uchida T, Kasai M, Oyama T, Suzuki T, Kobayashi Y, Watanabe T, Azuma T, Mori M, Terui Y, Yokoyama M, Mishima Y, Takahashi S, Ono C, Ohata J. Phase I study of inotuzumab ozogamicin (CMC-544) in Japanese patients with follicular lymphoma pretreated with rituximab-based therapy. Cancer Sci. 2010 Aug;101(8):1840-5. doi: 10.1111/j.1349-7006.2010.01601.x. Epub 2010 Apr 23. PMID 20491780
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3129K1-103